CLINICAL TRIAL: NCT04087850
Title: Encouraging Social Inclusiveness as a Means to Improving Academic Performance for Children at Risk Attention-Deficit/Hyperactivity Disorder (ADHD) and Typical Children
Brief Title: Encouraging Social Inclusiveness as a Means to Improving Academic Performance
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Responsible Party: Principal Investigator, Amori Yee Mikami, Professor, University of British Columbia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: R324A16005
Record Dates: First submitted 2019-09-06; First posted 2019-09-12 (Actual); Last update posted 2020-11-12 (Actual); Status verified 2020-11

CONDITIONS: ADHD
Keywords: peer relationships
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Some outcome measures are collected through interviewing children and their classmates, who would not be aware of the intervention condition of their classroom; this is because the intervention is delivered to the classroom teacher outside of class time.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Making Socially Accepting Inclusive Classrooms (MOSAIC) (Experimental)
  Interventions: Behavioral: Making Socially Accepting Inclusive Classrooms
- Typical Practice Control (No Intervention)

INTERVENTIONS:
Behavioral: Making Socially Accepting Inclusive Classrooms — Using a consultation model, study staff members met with teachers approximately twice per month and observed them an additional two times per month. The goal was to help teachers implement practices that create a socially accepting classroom climate for children.
  Arms: Making Socially Accepting Inclusive Classrooms (MOSAIC)

SUMMARY:
Children's peer relationships in elementary school are important to promote their academic learning and their social-emotional development. Many children with or at risk for Attention-Deficit/Hyperactivity Disorder (ADHD) have difficulty being accepted and getting along with their classroom peers. This study tested a classroom intervention that aimed to help improve the peer relationships of elementary school age children, with a particular focus on children with or at risk for ADHD.

ELIGIBILITY:
Inclusion Criteria:

-General education teachers of grades K-5 or children in these teachers' classrooms

Exclusion Criteria:

-None

Ages: 5 Years to 11 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 558 (Actual)
Dates: Start 2016-08-15 (Actual); Primary Completion 2019-07-01 (Actual); Study Completion 2020-07-01 (Actual)

PRIMARY OUTCOMES:
Children's Peer Relationships - Peer Report | Change from baseline to post-test (approximately 7 months after baseline)
  Assessed through peer sociometric interviews. The proportion of positive nominations, negative nominations, friendships, and the average liking rating received from peers will be calculated. More positive nominations and friendship nominations, fewer negative nominations, and higher liking ratings are considered to be positive outcomes.
Children's Peer Relationships - Child Self-Report | Change from baseline to post-test (approximately 7 months after baseline)
  Assessed through child self-report on the Classroom Life Measure. There are 9 items about peer relationships, each answered from a scale of 0-4. Scores range from 0-36 where higher numbers indicate more positive outcomes.
Children's Peer Relationships - Teacher Report | Change from baseline to post-test (approximately 7 months after baseline)
  Assessed through teacher report on the Dishion Social Acceptance Scale. The teacher estimates the proportion of classmates that like, dislike, and are neutral toward the child. Higher proportions of liking and lower proportions of disliking and neutrality represent positive outcomes.

SECONDARY OUTCOMES:
Children's Academic Functioning - Teacher Report | Change from baseline to post-test (approximately 7 months after baseline)
  Assessed through teacher report on the Academic Competence Evaluation Scales. This is a normed measure with 10 items about interpersonal skills, 8 about engagement, and 11 about motivation, each rated on a 1-5 scale. Each subscale represents the sum of the items on the subscale, and higher scores indicate positive outcomes.
Children's Academic Functioning - Teacher Report | Change from baseline to post-test (approximately 7 months after baseline)
  Assessed through teacher report on the Academic Performance Rating Scales. This is a 19 item scale with each item rated on a 1-5 metric. Some items are reverse scored. Higher scores indicate positive outcomes.
Children's Academic Functioning - Grades | Change from baseline to post-test (approximately 7 months after baseline)
  Assessed through grades on children's report cards. Higher grades indicates positive outcomes.
Children's Social Behaviors - Observations | Change from baseline to post-test (approximately 7 months after baseline)
  Assessed through behavioral observations on children's classroom behaviors. This is a proportion score indicating children's off-task, interfering, defiant, and verbally aggressive behaviors. Lower scores indicate positive outcomes.
Children's Social Behaviors - Observations | Change from baseline to post-test (approximately 7 months after baseline)
  Assessed through behavioral observations on messages written by children to one another, on codes representing the connection, support, and positivity in the messages children receive. Higher scores on these indicators and lower scores on indicators of platitudes indicate positive outcomes.
Children's Problem Behaviors - Teacher Report | Change from baseline to post-test (approximately 7 months after baseline)
  Assessed through teacher report of ADHD symptoms on the ADHD-4 Rating Scale. There are 18 symptom items, each rated on a scale of 0-3. Lower scores indicate positive outcomes.

CONTACTS AND LOCATIONS:
Overall Officials: Amori Mikami, PhD, Principal Investigator — University of British Columbia; Julie Owens, PhD, Principal Investigator — Ohio University

IPD SHARING:
Plan to Share IPD: No